CLINICAL TRIAL: NCT00360412
Title: A Multi-centre, Open Label Extension Study to Evaluate the Long-term Safety, Tolerability and Efficacy of E2007 as an Adjunctive Therapy in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Brief Title: A Study of E2007 as an Adjunctive Therapy in Levodopa Treated Parkinson's Disease Patients With Motor Fluctuations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to lack of efficacy.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-303; 2006-002339-26 (EudraCT Number)
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — perampanel

ARMS (1):
- E2007 (Experimental): During the first two weeks of the study, Patients received 1 x 2mg E2007 tablet. At the week 2 visit, patients who tolerated the 2 mg/day dose were up-titrated to receive 4mg/day (2 x 2 mg E2007 tablets). Patients not tolerating the 4 mg dose were allowed to down titrate to 2 mg. Patients who did not tolerate the 2 mg dose were withdrawn from the study. Patients returned at week 4, if their tolerance to the 4 mg/day dose was acceptable they remained on this dose for the maintenance phase of the study. If at any time their tolerance declined, they were to return for an unscheduled visit and the daily dose was reduced to 2 mg. If at any stage, 2 mg day wass not tolerated, the patient was withdrawn from the study.
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007

SUMMARY:
Patients who have completed one of the core trials (E2007-E044-301 or E2007-A001-302) and who meet inclusion/exclusion criteria will be enrolled and will enter the Titration Phase, lasting 4 weeks (weeks 0-3) followed by the Maintenance Phase, lasting 52 weeks (weeks 4-56). All patients will receive active study drug. During the Titration Phase, patients will receive E2007 2 mg once daily (o.d.) for 2 weeks followed by 4 mg o.d. for 2 weeks. During the Maintenance Phase, patients will receive 4 mg o.d. Patients not tolerating the study drug at 4 mg, will be allowed to down titrate to 2 mg. Patients not tolerating 2 mg will be withdrawn from the study.

Patients will have visits at 2, 4, 8, 20, 32, 44, and 56 weeks after study entry. In addition, a follow-up visit will occur 4 weeks after study treatment has ended (week 60).

A home diary will be completed in which patients rate themselves as either:

1. OFF
2. ON without dyskinesia
3. ON with non-troublesome dyskinesias
4. ON with troublesome dyskinesias
5. Asleep

These entries will be completed every half hour during the waking day and will be completed for 3 consecutive days following the visits at weeks 4, 8, 20, 32 and 44, and three days prior to the visits at weeks 56 and 60. At entry into the study (week 0) and at weeks 8, 20, 32, 44 and 56, the Unified Parkinson's Disease Rating Scale (UPDRS), Clinician's Global Impression of Change (CGIC) and Clinical Global Impression of Tolerance (CGIT) will be performed.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients with idiopathic PD who have fulfilled the entry criteria to either E2007-E044-301 or E2007-A001-302 and have completed that study up to and including the final efficacy visit. Patients will not be eligible if they withdrew from the core study prior to the final efficacy visit for any reason including lack of efficacy. Patients with SAEs which are ongoing or possibly or probably related to the study drug, will not be eligible for this study. Patients with ongoing adverse events categorized as severe and thought to be related to E2007 should not be entered. Patients with mild or moderate adverse events thought to be related to E2007 can be entered to the study if the investigator considers it safe.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Women of child bearing potential unless infertile (including surgically sterile) or practicing effective contraception (e.g., abstinence, IUD or barrier method plus hormonal method). These patients must have a negative serum or urine B-HCG test at their first study visit. These patients must also be willing to remain on their current form of contraception for the duration of the study. Postmenopausal women may be recruited but must be amenorrhoeic for at least 1 year to be considered of non-child bearing potential as determined by the investigator.
3. Patients with a past (within the past 5 years) or present history of drug or alcohol abuse as per DSM IV criteria.
4. Patients with a past (within one year) or present history of suicidal ideation or suicide attempts.
5. Patients with a past (within one year) or present history of psychotic symptoms requiring antipsychotic treatment. Patients may be taking anti-depressant medication, however the dose must be stable for 4 weeks prior to the baseline visit. Use of anti-psychotic medication including clozapine and quetiapine is prohibited even if the indication is for movement disorders.
6. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, gastro-intestinal, haematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.
7. Patients with significantly elevated liver enzymes (abnormal bilirubin or serum transaminase levels of more than 1.5 times the upper normal limit).
8. Medication known to induce the enzyme cytochrome P450 3A4 is prohibited throughout the study.
9. Current or prior treatment (within 4 weeks prior to entry visit) with tolcapone, methyldopa, budipine, reserpine, seroquel.
10. Patients with conditions affecting the peripheral or central sensory system unless related to Parkinson's disease (such as mild sensory or pain syndromes limited to OFF periods) that could interfere with the evaluation of any such symptoms caused by the study drug.
11. Patients receiving or with planned (next 12 months) deep brain stimulation.
12. Patients with any condition that would make the patient, in the opinion of the Investigator, unsuitable for the study.
13. Patients with clinically significant ECG abnormalities, including prolonged QTc (defined as QTc ≥ 450 msec).
14. Patients with previous stereotactic surgery (e.g., pallidotomy) for Parkinson's disease or with planned stereotactic surgery during the study period.
15. Patients on pergolide as of April 5, 2007.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 997 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (1):
- Philipps-University Marburg, Marburg, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel (Placebo During Core Study); Perampanel (Perampanel 2 mg or 4 mg During Core Study): Subjects entered this open-label extension study from the double-blind core studies (E2007-E044-301 and E2007-A001-302). Subjects started on perampanel 2mg once daily for two weeks, followed by 4mg once daily for 2 weeks (Titration Phase); Subjects then continued onto the maintenance phase of perampanel 4mg once daily for 2 weeks. Subjects that did not tolerate the study drug at 4mg were allowed to down-titrate to 2mg. Subjects that did not tolerate 2mg were withdrawn from the study.
Period: Overall Study
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Started | 333 | 664
Completed | 0 | 2
Not Completed | 333 | 662
Not completed — Adverse Event | 37 | 65
Not completed — Protocol Violation | 2 | 5
Not completed — Patient withdrew consent | 27 | 52
Not completed — Lack of therapeutic efficacy | 46 | 61
Not completed — Physician Decision | 2 | 4
Not completed — Other | 5 | 6
Not completed — Study termination by Sponsor | 214 | 469

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study) | Total
Number analyzed (Participants) | 333 | 664 | 997
Age, Customized [Number; unit: Participants] — Data comes from previous double-blind core studies (E2007-E044-301) and (E2007-A001-302).
  Participants
    <65 years | 187 | 357 | 544
    >=65 years | 146 | 307 | 453
Sex: Female, Male [Count of Participants; unit: Participants] — Data comes from previous double-blind core studies (E2007-E044-301 and E2007-A001-302). Safety Population - All subjects entering the open-label extension study who took at least 1 dose of perampanel
  Participants
    Female | 117 | 236 | 353
    Male | 216 | 428 | 644
Race/Ethnicity, Customized [Number; unit: Participants] — Data comes from previous double-blind core studies (E2007-E044-301 and E2007-A001-302). Safety population.
  Participants
    White | 320 | 643 | 963
    Black | 3 | 4 | 7
    Asian | 4 | 2 | 6
    Other | 6 | 15 | 21

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Daily OFF Time (Hours) During Open-label Extension Study
Description: OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 20, Week 32, Week 44, Week 56, Week 68
Population: Safety Population- all subjects entering the open-label extension study who took at least 1 dose of perampanel
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Number analyzed (Participants) | 333 | 664
Hours
  Week 0 | -0.78 (2.158) | -0.85 (2.498)
  Week 4 | -1.37 (2.483) | -1.16 (2.632)
  Week 8 | -1.21 (2.400) | -1.19 (2.568)
  Week 20 | -1.11 (2.537) | -1.34 (2.694)
  Week 32 | -0.91 (2.663) | -1.38 (2.676)
  Week 44 | -0.73 (2.371) | -1.44 (2.470)
  Week 56 | -0.64 (2.607) | -0.78 (2.010)
  week 68 | -0.92 (2.239) | -1.05 (1.820)

2. Secondary Outcome: Mean Change From Baseline in Total Daily ON Time (Without Dyskinesias or With Non-troublesome Dyskinesias) (Hours) During Open-label Extension Study
Description: ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor. This outcome measure was based on data collected through use of a patient diary.
Time Frame: Baseline, Week 0, Week 4, Week 8, Week 20, Week 32, Week 44, Week 56, Week 68
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Number analyzed (Participants) | 333 | 664
Hours
  Week 0 | 0.73 (2.389) | 0.65 (2.567)
  Week 4 | 1.02 (2.664) | 0.98 (2.665)
  Week 8 | 0.82 (2.741) | 0.96 (2.801)
  Week 20 | 0.95 (2.811) | 1.14 (2.803)
  Week 32 | 0.77 (2.716) | 1.05 (2.695)
  Week 44 | 0.60 (2.742) | 0.98 (2.634)
  Week 56 | 0.40 (2.596) | 0.02 (2.132)
  Week 68 | 0.50 (2.121) | 0.21 (1.539)

3. Secondary Outcome: Mean Change From Baseline in UPDRS Part II (ADL) Score in OFF State (Hours) During Open-label Extension Study
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part II assesses activities of daily living (ADL) based on 13 items, such as speech, hygiene, and falling. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms, for a range of total possible scores of 0-52. OFF state is when medication has worn off and is no longer providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 0, Week, 8, Week 20, Week 32, Week 44, Week 56, Week 68
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Number analyzed (Participants) | 333 | 664
Scores on a scale
  Week 0 | -0.36 (4.035) | -0.39 (4.567)
  Week 8 | -0.31 (4.752) | -0.60 (4.797)
  Week 20 | -0.38 (4.667) | -0.36 (5.152)
  Week 32 | 0.07 (5.018) | -0.12 (5.436)
  Week 44 | -0.22 (5.217) | -0.25 (5.390)
  Week 56 | -1.00 (5.228) | 0.38 (6.171)
  Week 68 | -3.00 (0) | 2.43 (5.623)

4. Secondary Outcome: Mean Change From Baseline in UPDRS Part III (Motor) Score in ON State (Hours) During Open- Label Extension Study
Description: Unified Parkinson's Disease Rating Scale (UPDRS) is a standardized assessment of the symptoms and signs of Parkinson's Disease. Part III assesses motor activity, based on 14 items, such as gait, facial expression, and rigidity. Participants receive a score of 0-4 points per item, with a higher score indicating more severe symptoms, for a range of total possible scores of 0-56. ON state is when medication is providing benefits with regard to stiffness, slowness, and tremor.
Time Frame: Baseline, Week 0, Week 8, Week 20, Week 32, Week 44, Week 56, Week 68
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Number analyzed (Participants) | 333 | 664
Scores on a scale
  Week 0 | -1.92 (6.945) | -1.87 (7.518)
  Week 8 | -3.17 (7.712) | -3.08 (8.273)
  Week 20 | -2.48 (7.425) | -2.72 (8.521)
  Week 32 | -2.86 (8.501) | -2.84 (7.677)
  Week 44 | -2.23 (8.428) | -2.07 (9.209)
  Week 56 | -1.91 (7.770) | -0.84 (9.428)
  Week 68 | -7.00 (0) | -1.29 (6.775)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were defined as treatment emergent in this study if the start date of the event was on or after the start of study medication in this study. Adverse events that occurred 30 days after the last dose of study drug were 'post-treatment'.
Arm/Group | Perampanel (Placebo During Core Study) | Perampanel (Perampanel 2 mg or 4 mg During Core Study)
Serious Adverse Events (participants affected / at risk) | 33/333 | 57/664
Other Adverse Events (participants affected / at risk) | 104/333 | 201/664
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=333) | Perampanel (Perampanel 2 mg or 4 mg During Core Study) (N=664)
Parkinson's disease (Nervous system disorders) | 1 | 4
On and off phenomenon (Nervous system disorders) | 1 | 2
Akinesia (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 0 | 1
Bradykinesia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Hyperkinesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 2
Acute Psychosis (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Pathological gambling (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicidal attempt (Psychiatric disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Abdomina strangulated hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Hematemesis (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (Placebo During Core Study) (N=333) | Perampanel (Perampanel 2 mg or 4 mg During Core Study) (N=664)
Fall (Injury, poisoning and procedural complications) | 24 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 35
Dyskinesia (Nervous system disorders) | 33 | 72
On and off phenomenon (Nervous system disorders) | 42 | 73
Somnolence (Nervous system disorders) | 22 | 33
Insomnia (Psychiatric disorders) | 17 | 37

LIMITATIONS AND CAVEATS:
Due to early termination, a limited number of subjects (only 2) completed this open-label extension study. The majority of subjects did not reach the scheduled Week 56 assessment. Many outcomes could only be analyzed to Week 68 as a result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No